CLINICAL TRIAL: NCT01002417
Title: An Adaptive, Phase 2b/3, Double-Blind, Randomized, Placebo-Controlled Study to Establish the Dosage, Efficacy, and Safety of MCS-2 in Treating Lower Urinary Tract Symptoms Suggestive of BPH in Treatment-Naive Male Subjects
Brief Title: MCS in the Treatment of Lower Urinary Tract Symptoms
Acronym: MCS_LUTS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Health Ever Bio-Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCS-2-US-a
Record Dates: First submitted 2009-10-25; First posted 2009-10-27 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; Multi-carotenoids; MCS-2; Lower Urinary Tract Symptoms; International prostate symptom scores
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Both the phase 2b and phase 3 parts of the study have the placebo arm.
  Interventions: Drug: Placebo
- MCS-2 15 mg/day (Active Comparator): For the phase 2b part of the study. It can also be used in the phase 3 part of the study if MCS-2 15 mg/day is selected as the optimal dosage.
  Interventions: Drug: MCS-2 15 mg/day; Drug: MCS-2 30 mg/day
- MCS-2 30 mg/day (Active Comparator): For the phase 2b part of the study. It can also be used in the phase 3 part of the study if MCS-2 30 mg/day is selected as the optimal dosage.
  Interventions: Drug: MCS-2 15 mg/day; Drug: MCS-2 30 mg/day

INTERVENTIONS:
Drug: MCS-2 15 mg/day — One MCS-2 15 mg soft-gel capsule plus one matching placebo capsule, oral daily for 12 weeks.
  Other Names: MUS
  Arms: MCS-2 15 mg/day; MCS-2 30 mg/day
Drug: MCS-2 30 mg/day — Two MCS-2 soft-gel capsules, oral daily for 12 weeks.
  Other Names: MUS
  Arms: MCS-2 15 mg/day; MCS-2 30 mg/day
Drug: Placebo — Two matching placebo soft-gel capsules, oral daily for 12 weeks.
  Other Names: MCS matching placebo
  Arms: Placebo

SUMMARY:
The hypothesis of the study is to examine whether MCS-2 is safe and effective in the treatment of lower urinary tract symptoms suggestive of benign prostatic hyperplasia.

DETAILED DESCRIPTION:
This is an adaptive trial design, that combines elements of a Phase 2b (dose ranging) study and a Phase 3 (hypothesis testing) study, the objectives for the two phases are separate.

Phase 2b Objectives: The primary objective of the Phase 2b portion of this study is to evaluate, in a treatment-naïve population, the 0 mg (placebo), 15 mg, and 30 mg MCS-2 in terms of dose response and to determine the optimal dose to be used in the Phase 3 portion of this trial. The secondary objective of this portion of the study is to evaluate the safety and tolerability of the 15 mg and 30 mg MCS-2.

Phase 3 Objectives: The primary objective of the Phase 3 portion of this study is to evaluate, in a treatment-naïve population, the effectiveness of the MCS-2 (at the dosage determined in the Phase 2b portion of this study), as compared to MCS placebo (0 mg), in reducing the lower urinary tract symptoms (LUTS) suggestive of benign prostatic hyperplasia (BPH). The secondary objective of this study is to evaluate the safety and tolerability of MCS-2 (at the dosage determined in the Phase 2b portion of this study), as compared to MCS placebo (0 mg).

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 40 years old
* Not being treated for BPH or LUTS
* PSA ≦ 4 ng/ml and no pathologically-proven prostate cancer
* I-PSS ≥ 10
* No known malignancy
* AST/ALT ≦ 3X UNL
* Creatinine ≦ 3X UNL
* Subjects who sign the informed consent form

Exclusion Criteria:

* Subjects' LUTS are not BPH-related
* Have been treated with pelvis irradiation or pelvic surgery
* Plan to undergo any invasive procedures within the study period
* Active infection or inflammation
* Considered ineligible by the investigators

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2010-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in International Prostate Symptom Scores | 12 weeks

SECONDARY OUTCOMES:
Changes in I-PSS subscores | 12 weeks
Changes in I-PSS QOL index | 12 weeks
Changes in urine flow rate | 12 weels
Incidence of treatment-emergent adverse events (TEAE) | 12 weeks
Incidence of withdrawals due to TEAEs | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allan J Pantuck, MD, MS, FACS, Principal Investigator — University of California, Los Angeles
Locations (1):
- David Geffen School of Medicine at UCLA, Los Angeles, California, United States